CLINICAL TRIAL: NCT03568773
Title: Influence of Polymorphysms in the Fto and Ppar Gen Genes, Systemic Inflammation and Oxidative Stress in the Magnitude of Weight Loss Induced by Intermittent or Moderate Continuous High Intensity Training Programs
Brief Title: Influence of Genetic and Physiological in Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Raquel Suelen Brito da Silva, Master/ Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUP
Record Dates: First submitted 2018-05-03; First posted 2018-06-26 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Overweight and Obesity; Chronic Disease
MeSH Terms: conditions — Overweight; Obesity; Chronic Disease | interventions — High-Intensity Interval Training; Control Groups

STUDY DESIGN:
Intervention Model Description: Experimental, controlled and randomized study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (Experimental): The HIIT protocol is being performed with the cycling mode. The program consists of repeated intense explosions alternating with recovery intervals.
  The adaptation period consists of 4 shots of 20 seconds interspersed by 180 seconds interval (active recovery). From the first to the fourth week the volunteers performed from four to six race shots from 30 to 45s with intervals from 180s to 120s. From the fifth week until the end of the intervention, training takes place with six shots of 60s with a 120s interval between running shots. The work intensity for all sessions is above 95% of VO2max, with 30W of recovery. In addition, participants refer to number 19 on the Borg Scale. Sessions range from 12 to 36 minutes without heating and recovery. In total there are 12 weeks of training.
  Interventions: Other: High-intensity interval training
- Aerobic exercise moderate intensity (Experimental): The training protocol was started, with the sessions held in the open air. From the first to the fourth week, the volunteers gave sessions of 40 to 60 minutes, intensity in L1, three sessions / week. In the fifth week, the intensity was increased to the midpoint between L1 and half of L2, maintaining 60 minutes per session and frequency three times per week. From the sixth week, the weekly frequency increased to five days, with three supervised sessions and two unsupervised sessions, but with a smartphone application that recorded distance traveled and intensity. From the ninth week on, the weekly frequency was maintained and the intensity increased for L2. In supervised sessions, training intensity is also monitored by heart rate using a Polar heart rate monitor.
  Interventions: Other: Aerobic exercise moderate intensity
- Control Group (Experimental): The control group attends stretching classes once a week and sessions lasting 60 minutes. At the end of the fifteen weeks (three weeks of adaptation and twelve weeks of training) of the study, these volunteers will be invited to engage in the aerobic training program regardless of their participation in the research.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: High-intensity interval training — HIIT training is being conducted on a three-day weekly frequency on a stationary bike. The protocol consisted of two weeks of adaptation with 12 weeks of training that alternated between sprints ranging from 30 s to 60 s (> 95% VO2max), and active recovery ranging from 180 s to 120 s (30 W on the bicycle).
  Arms: High-intensity interval training
Other: Aerobic exercise moderate intensity — The aerobic training is performed in a walking or running mode, with three weeks of adaptation (2x / wk - 20 to 30 minutes / session, <threshold 1) and 12 weeks of training (3 to 5x / wk - 40 to 60 minutes / session, with prescribed intensities between the anaerobic threshold - L1 and the respiratory compensation point - L2).
  Arms: Aerobic exercise moderate intensity
Other: Control Group — The control group is participating in lengthening classes to increase the adherence and control of the influencing variables. Classes are being held once a week for 60 minutes.
  Arms: Control Group

SUMMARY:
The study focuses on the influence of polymorphism in the FTO genes rs9939609 and PPARᵧ Pro12Ala, oxidative stress and systemic inflammation on changes in body composition and rest metabolism induced by HIIT and continuous aerobic programs in obese or overweight individuals.

DETAILED DESCRIPTION:
Although the positive effects of continuous aerobic training are already well documented in the literature on health aspects. The weight loss induced by physical training is still very discrete when compared to other antiobesity means. Studies demonstrate an important variability in responses to physical exercise, indicating that individuals respond more or less to weight loss. Among these aspects, the factors that may influence exercise-induced weight loss have not yet been elucidated. Thus, the objective of the study is to analyze the influence of polymorphism in the genes FTO rs9939609 and PPARᵧ Pro12Ala, oxidative stress and systemic inflammation on changes in body composition and rest metabolism induced by continuous and continuous aerobic programs. Healthy individuals with overweight and / or obesity, aged 20-45 years, were randomly assigned to three groups: Continuous Aerobic (AC), Intermittent High Intensity Training (HIIT) and Control Group (CG). Groups (AC) and (HIIT) engaged in a 12-week program. Before the start of the program, at the sixth week and 48 hours after the intervention, they performed blood collections, ergospirometry, dual X-ray densitometry (DEXA), nutritional assessments. In addition, collection of buccal mucosa was performed for genotyping of polymorphisms studied. Initial differences between the groups, as well as between the dependent variables studied will be assessed using the two-way ANOVA test or its non-parametric equivalent. Correlation and regression tests will be performed to verify the influence of the independent variables and the magnitude of the exercise-induced weight loss, according to the normality of the data or differences between the standard deviations. The hypothesis tested is that genetic and physiological factors influence the weight loss independent of the training modality.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 20-45 years;

Were insufficiently active for at least six months prior to recruitment as determined by the International Physical Activity Questionnaire (IPAQ) (<150 minutes of moderate to intense physical activity / week) (MATSUDO, 2001);

Were overweight or obese (BMI between 25kg / m2 and 39.9kg / m2) (WHO, 2015);

Did not suffer any change in weight (more than 5kg in the last three months);

Do not be smokers or acololistas (maximum of 2 doses / day);

They may not be users of supplements and / or medications that influence weight loss or weight gain;

No history of coronary, respiratory, metabolic, or musculoskeletal disease affecting ability to participate in the training program;

Have been considered fit in an exercise test performed immediately prior to physical intervention;

Women are not menopausal (menstrual cycle stopped more than one year) or have symptoms related to the climacteric phase.

Exclusion Criteria:

Individuals who lack at least 25% of the total training program or two consecutive weeks;

Initiate medication treatment, supplementation, diet and / or other physical training program during the intervention period;

During training, osseous and / or myoarticular lesions that affect the ability to continue participating in the intervention.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2016-03-10 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Body Composition. The changes are being evaluated. | Before the intervention protocol and 48 hours immediately after the last exercise session.
  The procedure used for analysis is done using a Dual Energy Radiological Absortiometry (DEXA) equipment. The measurement of the body fat and fat free mass percentage measure is obtained by means of a full body scan using the LUNAR PRODIGY DF + 14.319 Radiation (Madison, WI) brand device, following manufacturer's protocols. The body mass is evaluated by means of a balance (Sanny®, São Bernardo do Campo - São Paulo, Brazil), with the volunteer barefoot and in orthostatic position using a Toledo scale sensitive to 100 g. The stature is evaluated by a stadiometer with a tape calibrated at 0.1 of the same mark. Waist circumference and other body perimeters are measured with a 0.1 cm Anthropometric Tape (Sanny®, São Bernardo do Campo - São Paulo, Brazil). Weight and height data are used to calculate BMI using the equation adopted by the WHO: BMI = (Weight / (Stature) 2).

SECONDARY OUTCOMES:
Metabolic Rate of Rest. The changes are being evaluated. | Before the intervention protocol and 48 hours immediately after the last exercise session.
  The metabolic rate was measured using a gas spirometry analyzer. After having fasted from 8:00 pm the previous day, the volunteers were referred to the laboratory shortly after the awakening and were invited to remain seated in a thermoneutral environment for 30 minutes. For the next 30 minutes, VO2, VCO2, VE and RER were monitored until variations of no more than 10% occurred when five-minute intervals were compared. Once this steady state was obtained, these variables were recorded for five minutes. The calculation of the resting metabolic rate is done according to Macdonald (1990).
Lipid and Glycemic Profile. The changes are being evaluated. | The collections will be done 24 hours before, in the 6th week and 48 hours after the end of the intervention.
  Collections of 10 ml of blood from the antecubital vein will be performed early in the morning, with fasting from 10 to 12 hours. The collections will be done 24 hours before, in the 6th week and after the intervention period. They will remain seated for 10 minutes for subsequent collection. Five milliliters of blood will be placed in EDTA-containing test tubes, protected from light and gently homogenized by inversion. The other 5ml will be placed in tubes without anticoagulants. They will then be centrifuged at 3,000 rpm for 10 min. The plasma or serum will be separated, placed in eppendorf tubes and refrigerated at -20 ° C until analysis. All analyzes will be carried out using a commercial kit of the Labtest brand (Minas Gerais-Brazil). The analyzes will be carried out on serum samples using commercial Labtest kits (Minas Gerais, Brazil), following the manufacturer's recommendations and on a Labmax 240 premium automatic analyzer (Lagoa Santa-MG, Brazil).
Oxidative stress (Malondialdehyde). The changes are being evaluated. | The collections will be done 24 hours before, in the 6th week and 48 hours after the end of the intervention.
  10 ml of blood will be collected in the beginning of the morning, with fasting of 10 to 12 hours, being done 24 hours before, in the 6th week and after the intervention period. Five milliliters of blood will be placed in test tubes containing EDTA and protected from light and the other 5ml will be placed in tubes without anticoagulants and centrifuged at 3,000 rpm for 10 min. The plasma or serum will be separated, placed in eppendorf tubes and refrigerated at -20 ° C until analyzed by a commercial kit of the Labtest brand (Minas Gerais, Brazil). For this, 250 μl of sample will be added to KCl and incubated in a water bath (37 ° / 60 minutes). The mixture will be precipitated with 35% AA perchloric acid and centrifuged at 14,000 rpm for 10 minutes at 4 ° C. The supernatant will be transferred to eppendorfs and 400μl of 0.6% thiobarbituric acid is added and incubated at 95-100 ° C for 30minutes. The material will be read in a spectrophotometer at a wavelength of 532nm.
Oxidative stress (Total antioxidant capacity). The changes are being evaluated. | The collections will be done 24 hours before, in the 6th week and 48 hours after the end of the intervention.
  10 ml of blood will be collected in the beginning of the morning, with fasting of 10 to 12 hours, being done 24 hours before, in the 6th week and after the intervention period. Five milliliters of blood will be placed in test tubes containing EDTA and protected from light and the other 5ml will be placed in tubes without anticoagulants and centrifuged at 3,000 rpm for 10 min. The plasma or serum will be separated, placed in eppendorf tubes and refrigerated at -20 ° C until analyzed by a commercial kit of the Labtest brand (Minas Gerais, Brazil). The evaluation of the total antioxidant capacity will be performed through DPPH. For analysis, 100 μl of plasma will be added to 3.9 ml of vortexed DPPH solution, set to stand for 30 minutes and then centrifuged at 10,000 rpm for 15 minutes at 20 ° C. The supernatant will be used for spectrophotometer reading at 515 nm wavelength, using distilled white water. The result will be expressed as a percentage of antioxidant activity.
Systemic Inflammation (Plasma ultra-sensitive C-reactive protein). The changes are being evaluated. | The collections will be done 24 hours before, in the 6th week and 48 hours after the end of the intervention.
  10 ml of blood will be collected in the beginning of the morning, with fasting of 10 to 12 hours, being done 24 hours before, in the 6th week and after the intervention period. Five milliliters of blood will be placed in test tubes containing EDTA and protected from light and the other 5ml will be placed in tubes without anticoagulants and centrifuged at 3,000 rpm for 10 min. The plasma or serum will be separated, placed in eppendorf tubes and refrigerated at -20 ° C until analyzed by a commercial kit of the Labtest brand (Minas Gerais, Brazil). The concentration of hs-CRP will be quantified by immunoturbidimetry in serum samples. Calibration will use the Calibra Calibrator from Labtest (Calibra Plus PCR-ultra - Ref-345). Absorbance will be obtained on the Labmax 240 premium automatic analyzer at 540 nm wavelength. The concentrations of hs-CRP will be determined by the commercial kit (Labtest, Minas Gerais, Brazil) according to the manufacturer's instructions.
Systemic Inflammation (Analysis of alpha-1-glycoprotein acid). The changes are being evaluated. | The collections will be done 24 hours before, in the 6th week and 48 hours after the end of the intervention.
  10 ml of blood will be collected in the beginning of the morning, with fasting of 10 to 12 hours, being done 24 hours before, in the 6th week and after the intervention period. Five milliliters of blood will be placed in test tubes containing EDTA and protected from light and the other 5ml will be placed in tubes without anticoagulants and centrifuged at 3,000 rpm for 10 min. The plasma or serum will be separated, placed in eppendorf tubes and refrigerated at -20 ° C until analyzed by a commercial kit of the Labtest brand (Minas Gerais, Brazil). The A1GPA concentration will be quantified by immunoturbidimetry using the commercial kit (Labtest, Minas Gerais, Brazil) as per manufacturer's instructions. Calibration will use the Calibra Calibrator from Labtest (Calibra Plus Protein - Ref-346). The absorbance will be obtained in the Labmax 240 premium automatic analyzer (Lagoa Santa-MG, Brazil), at wavelength 340nm.
DNA Extraction and Genotyping | The genetic collection will be made in the 6th week of the intervention.
  Oral cell samples were collected through a mouthwash for 60 seconds of 5 ml of 3% sucrose solution. The resulting contents of the mouthwash were transferred to a 15 ml tube, which immediately afterwards was placed in a solution of TNE (17 mM Tris-HCl pH 8.0, 50 mM NaCl and 7 mM EDTA), diluted to 66% alcohol and autoclaved distilled water.After this, the extraction and genotyping process followed the recommendations of Saiki et al. (1985)

IPD SHARING:
Plan to Share IPD: No